## **COVER PAGE**

Effects of Cranial Electrotherapy Stimulation on Psychological Distress and Maternal Functioning in New Mothers during the Postpartum Period

NCT03210155

Research protocol/IRB

07.01.20

| ORC USE ONLY | |
|--------------|--------|
| HSRP #: | |
| Date Rec | eived: |

# Human Subjects Research Protocol for Exempt, Expedited, or Full Board Review



| Instructions and Researcher | Certifications | Failure to follow ma | v result in a dela | v in processing |
|---|---|---|---|---|

Complete this form if "research" will be conducted.

Do not complete this form for:

- 1. non-research activities; or
- 2. to fulfill TAMUCC coursework only without a research activity or element.

By signing this Human Subjects Research Protocol for Exempt, Expedited, or Full Board Review (HSRP), all Principal Investigators (PIs), co-PIs, and personnel (collectively, "Researchers") certify the following:

- 1. CITI Training "Human Subjects Basic Refresher Course" has been completed and is current for **any research activity** regardless of source of funding or whether unfunded (expires after three years);
- 2. CITI Training "Responsible Conduct of Research Course" has been completed and is current <u>only if</u> the source of funding is the <u>National Institutes of Health (NIH)</u> or the <u>National Science Foundation (NSF)</u> (expires after three years);
- 3. Have read and understood the responsibilities set forth in TAMUCC Rule 15.99.01.C1.01;
- 4. Have read and reviewed this HSRP; any applicable supporting documentation or third-party approval has been obtained from the appropriate authority and has been included as an attachment to the HSRP (e.g., recruitment script, informed consent, parental consent, child assent, public school district approval, facility use permission, grant, Translator Certification, Interpreter Certification, etc); have signed the HSRP electronically;
- 5. Will immediately report any adverse event to either the Institutional Review Board (IRB) or the Research Compliance and Export Control Officer:
- 6. Have submitted the HSRP a minimum of thirty (30) days in advance of the anticipated start date (additional time is required for review at full board); will communicate whether there is a firm start date or other deadline associated with the HSRP;
- 7. If the HSRP is submitted for a doctoral dissertation, have coordinated with the College of Graduate Studies (CGS) to meet its requirements; and
- 8. Will submit a Completion Report at the conclusion of research under this HSRP.

After completing the foregoing, submit the HSRP with supporting documentation via email to the IRB Mailbox: irb@tamucc.edu

#### For questions, email:

Dr. Edward Orona, Research Compliance Coordinator, edward.orona@tamucc.edu

Caroline Lutz, JD, Research Compliance and Export Control Officer, caroline.lutz@tamucc.edu

Researchers

| | Name | Emai<br>(use TAMUC | | | College | Category | Categ<br>(Oth | |
|---|---|---|---|---|---|---|---|---|
| PI | R | | 18.8.1 | Dec , i'' ii | Nursing & Health Sciences | Other | | |
| Co-PI (1) | | and Lui | | | 00022, | | | 25.7 |
| Co-PI (2) | 791813<br>7 17 1 1 | | | | | | | |
| Co-PI (3) | | | | | | | | |
| Co-PI (4) | 4 | | | | | | | |
| Co-PI (5) | | | | | | | | |
| Overvie | :w | | | | J[L | W. SEMENTAL | | 975 375 |
| <b>A.</b> Resear | ch Classification: Research Pro | ject | | | Other: N/A | | | 3111 |
| For guidan | ce, see Determination of Level of Re | view at the end of the | e HSRP. | 1 | | | | |
| <b>B.</b> Level o | f Review: Expedite | d (1) | v- | | the of the same | 21 (20 12 | | |
| <b>C.</b> Indicate funding ap | e whether external No | Award St | tart N/ | A | Maestro #: N | /A | | |
| <b>D.</b> Title: | Effects of Cranial Electroduring the Postpartum I | | ion on | Psych | ological Distress and Mate | rnal Functioning in New | Mother | rs |
| E. Researd<br>Anticipate<br>Start Date | ed Upon IRB approval. | | | F. Est | timated Completion Date: | | | |
| Purpose | e and Objective | 1.3. <b>1</b> 3.0128671 (1 | | | esa sur danna lavor que | | | |
| A. Descri | be the purpose of the research | in layman's term | <b>S.</b> | | gel | | | |
| | oose of this study is to evaluate in functioning in first time new m | | | | erapy stimulation (CES) on | anxiety, insomnia, depre | ession, a | and |
| B. Descri | be the objective(s) and/or rese | arch questions <u>in</u> | layma | n's te | rms. | 3 | | |
| following<br>effect of (<br>Anxiety F | nary objective of this study is to<br>g childbirth. The secondary obje<br>CES on maternal functioning in<br>Rating Scale (HAM-A14) perforn<br>at for detailed information relat | ectives are to: (1) on<br>new mothers follon<br>well as a screen | determ<br>wing | ine th | e effects of CES on depress<br>irth, and (3) to examine if i | sion and insomnia; (2) exitems 1 & 2 on the 14 item | xplore th<br>m Hami | he |
| Particip | oants; Recruitment | | | | | an Salebarah ada mat | | |
| Participa | ants | | | | | | | |
| <b>A.</b> Indicate<br>answered | e whether the following popula | tions will be speci | fically | target | ed for inclusion in the rese | earch. Each category mus | st be | |
| Adults ove | er the age of 18 (able to legally | consent) | Y 🖂 | Ν□ | Prisoners (adults or juven | iles) | Y 🗀 | N⊠ |
| Adults ove | er the age of 18 ( <u>unable</u> to lega | lly consent) | Y 🗀 | N⊠ | Participants whose first la | nguage is <u>not</u> English | Y 🗀 | N⊠ |

| Minors under the age of 18 | Y 🗀 | N 🖂 | Students enrolled in a researcher's course(s) | Y 🗀 | N⊠ |
|---|---|---|---|---|---|
| Pregnant Women, fetuses, and/or neonates Note: Projects including this vulnerable population are <i>generally</i> health care/ medical studies specifically targeting research of pregnant women, fetuses, and/or neonates. Pregnant women can be included in projects if all inclusion criteria is met and a specific exclusion is not part of the project design. Select "No" unless the project specifically involves the inclusion of pregnant women, fetuses, and/or neonates. | | | Employees under the direct supervision of a researcher | Y 🗀 | N⊠ |

**B.** Describe the criteria to determine who is included or excluded in the final participant population (e.g., minimum age, grade range, physical characteristics, learning characteristics, professional criteria, etc).

Instruments: See attached document entitled "Instrument Description" for detailed information related to this the scales referenced in this protocol.

The Hamilton Anxiety Rating Scale (HAM-A14)

Hamilton Depression Rating Scale17 (HAM-D17)

The Pittsburgh Sleep Quality Index (PSQI19)

The Insomnia Severity Index (ISI7)

The Barkin Index of Maternal Functions (BIMF20)

### Screening and Inclusion Criteria:

- 1. Participant must have a total score of  $\geq$  16 on the HAM-A14 and  $\geq$ 2 on both Hamilton Anxiety Rating Scale (HAM-A14) item 1 (anxious mood) and item 2 (tension) at screening and baseline [74] to be considered for inclusion into the study.
- 2. Participant is a primiparous new mother, 18-45 years inclusive, who had an uncomplicated vaginal or cesarean birth, gave birth to a healthy baby and both mother and baby are healthy at enrollment and randomization in the study.
- 3. Sexually active female participants of childbearing potential must be self-report practicing, at least, one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female participants of childbearing potential must have a negative urine pregnancy test before receiving study treatment.
- 4. Written informed consent must be obtained from the participant before study participation.
- 5. Participant is in good medical health.
- 6. No current abuse of alcohol or other substance.
- 7. Capable of giving informed consent.
- 8. Capable of doing active or sham CES treatments and completing all study requirements independently
- 9. For compliance, participants need to have completed 85% (36) of treatments to continue participation in the study

#### **Exclusion Criteria:**

- 1. Participant had complications during or after a vaginal or cesarean delivery.
- 2. Participant had multiple births.
- 3. Participant meets DSM-V criteria for a mental disorder diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by medical history and/or self-report.
- 4. Participant is clinically judged by the investigator to be at risk for suicide or is acutely suicidal. Participant has attempted suicide one or more times within the past twelve months.
- 5. Participant has a Hamilton Anxiety Rating Scale (HAM-A14) score above 30 which suggests a very severe clinical level of anxiety symptoms.
- 6. Participant has a Hamilton Depression Rating Scale (HAM-D17) score above 30 which suggests a very severe clinical level of depressive symptoms.
- 7. Participant has a psychiatric condition that would require inpatient or partial psychiatric hospitalization.
- 8. Participant has a significant history of medical disease (i.e. cardiovascular, hepatic (e.g., cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological (seizures), gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
- 9. Participant is pregnant, planning to become pregnant. If a participant becomes pregnant, she will be dropped from the study immediately and followed appropriately.
- 10. Participant has had concomitant therapy with another investigational drug, or participation in an investigational drug study within one month before entering this study.
- 11. Participant has a history of poor compliance or in the Investigator's judgment any participant who is not compliant with the requirements of the study.
- 12. Participant has had previous trial of CES.

C. Target number of participants (use a minimum target if a specific target is not appropriate for the research design).

A power analysis indicated that 44 (22 participants in treatment group and 22 participants in sham group + 5 (10% for attrition) = 49 participants and would be the minimum needed for this study. Therefore, to account for possible attrition, I will recruit at total of 50 participants (25 subjects in treatment group and 25 subjects in sham group).

#### D. Non-TAMUCC Participants or Facility

Complete this section <u>only if</u> the research will be conducted at a third-party facility <u>or</u> participants will be recruited from a third-party site (non-TAMUCC).

Provide the non-TAMUCC location or non-TAMUCC participants to be recruited here (include any permission as an attachment).

Two OB/GYN clinics have agreed to let the Principal Investigator (PI) to recruit participants from their clinics. Letters of support are attached.

R

#### Recruitment

**E(1). Method.** Describe methods that will be used to identify the potential participants.

The PI or Research Assistant (RA) will recruit potential participants. Healthy primiparous new mothers in the postpartum period (defined as one year after childbirth) with uncomplicated vaginal or cesarean deliveries who gave birth to healthy infants and have a healthy infant at enrollment in the study. To enroll in the study, participants must score  $\geq$ 2 on both HAM-A14 item 1 (anxious mood) and item 2 (tension) and have a total score of  $\geq$  16 on the HAM-A14 at baseline. I included participants with lower HAM-A14 scores than is typically used in generalized anxiety disorder (GAD) clinical trials (i.e., HAM-A14 >20) since the participants included will be a "healthy" population. Using this approach will also improve the generalizability of results to clinical practice.

**E(2). Materials.** Describe how potential participants will be recruited, what materials will be used (include as an attachment), and how they will be distributed (i.e., who, what, when, where, and how).

Instruments: See attached document entitled "Instrument Description" for detailed information related to this the scales referenced in this protocol.

The Hamilton Anxiety Rating Scale (HAM-A14)

Hamilton Depression Rating Scale17 (HAM-D17) The Pittsburgh Sleep Quality Index (PSQI19)

The Insomnia Severity Index (ISI7)

The Barkin Index of Maternal Functions (BIMF20)

Recruitment and data collection is designed to fit into routine clinic procedures and scheduling and will be conducted in collaboration with clinic staff, administrators, and healthcare providers. Recruitment fliers briefly describing the study will be distributed by clinic staff in designated areas of the clinic. The PI or RA will conduct an information and training session with clinic staff. Potential participants who had uncomplicated vaginal or cesarean deliveries and healthy newborns will be told about the study by the clinic staff or health care provider.

If the new mother indicates interest in participating in the study, she will be asked to complete the background and demographic form and screening form (HAM-A14 item 1 (anxious mood) and item 2 (tension). The clinic staff member will place the potential participant's completed materials in a sealed envelope and place in a locked file cabinet in an inner-clinic office within the clinic to be picked by the PI or RA weekly. The PI or RA will review the background and demographic form, screen the participant's responses against the inclusion/exclusion criteria, and review results of screening form. To enroll in the study, participants must score  $\geq$ 2 on both HAM-A14 item 1 (anxious mood) and item 2 (tension) at screening and have a total score of  $\geq$  16 on the HAM-A14 at baseline. I included subjects with lower HAM-A14 scores than is typically used in GAD clinical trials (i.e. HAM-A14 >20) since the subjects included will be a "healthy" population.

The potential participant will be notified by the PI or RA if she qualifies for the study or does not meet the criteria for the study. If a new mother qualifies for the study, the PI or RA will briefly describe the study and time commitment. The PI or RA will explain the study's purpose and procedures and read the consent form to all potential participants. After the potential participant's questions are addressed and verbal consent to participate is obtained, the new mother will sign the informed consent form. If the new mother agrees to participate, an appointment will be scheduled at the participants' next scheduled clinic visit or at the current time and location with the PI or RA to complete Visit 1. Participants may also choose to complete study visits 1-3 during their current visit or at another designated location with the PI.

| <br>· · |
|---------|

E(3). Incentives. If applicable, provide the amount, type, and time of distribution of any payment/incentive to participants.

All participants have the opportunity to receive a total of \$100.00 to compensate for their time:

Visit 1: \$40.00 Visit 2: \$20.00 Visit 3: \$40.00

## Identification of Participants; Data Collection and Storage; Equipment; Records Retention

**A. Identification of Participants.** Indicate whether the data collected may contain individual identifiers (need for "confidentiality"), or whether the data will be collected anonymously.

#### Confidential

**B. Data Collection.** Describe the method(s) or procedure(s) for data collection <u>in step-by-step, layman's terms</u> (include collecting party, frequency, duration, location, etc).

The use of audio or video recording must be justified by the research purpose/objective or future research.

Participants will complete a daily 60 minute CES treatment and meet with the PI for three visits three weeks apart for a total of six weeks. Each visit will take approximately 60-80 minutes to complete.

#### • Visit 1/First day of treatment

During study Visit 1 the PI or RA will explain the study and answer any questions. Participants will complete a urine pregnancy test. If the urine pregnancy test is negative baseline measures using the HAM-A14, HAM-D17, PSQI19, ISI7, and BIMF20 questionnaires will be completed by the participant with researcher assistance. Participants will then be given an Alpha-Stim® AID CES device kit with a serial number. The PI or RA will instruct participants on how to use the Alpha-Stim® AID CES device; then the participant will be asked to complete a 60-minute treatment. After the completion of the treatment, the participant will be asked about any side-effects or problems the participant many have experienced. Any side-effects information will be recorded on a side-effect form using the subject's words that describe what happened. The protocol for study treatments at home will be explained to you, and any questions will be answered. The participant will be reminded to complete your daily 60 minute CES treatment before the Visit 2 meeting. The participant will receive a \$40.00 Target Gift Card after Visit 1.

#### • Visit 2

At study Visit 2 The participant will be asked to complete a urine pregnancy test. If the urine pregnancy test is negative the participant will be asked to complete the HAM-A14, HAM-D17, PSQI19, ISI7, and BIMF20 questionnaires with researcher assistance. Your log will be reviewed and discussed. The participant will be asked about any side-effects that the participant may have experienced. The protocol for study treatments at home will be reviewed and the following device supplies will be given to you: six new AAA batteries and two 15ml. bottle conducting solution. The process of how to contact the PI or RA will be reviewed. The participant will be reminded to complete your daily 60 minute CES treatment before the Visit 3 meeting. The participant will receive a \$20.00 Target Gift Card after Visit 2.

#### Visit 3/ Last day of treatment

At study Visit 3 The participant will be asked to complete a urine pregnancy test. If the urine pregnancy test is negative the participant will be asked to complete the HAM-A14, HAM-D17, PSQI19, ISI7, and BIMF20 questionnaires with PI or RA assistance. The subject's log will be reviewed and discussed as needed. The participant will be asked about any side–effects that the participant may have experienced. The Alpha-Stim® AID CES device and all supplies will be returned to the study team. The participant will receive a \$40.00 Target Gift Card after Visit 3.

**C. Equipment.** Describe any equipment to be used (e.g., audio, visual), ownership (e.g., TAMUCC, personal), and methods of storage (e.g., password, location).

Study Device: The Alpha-Stim® AID will be used for this study (Figure 1). The Alpha-Stim® AID is a prescriptive device and is FDA cleared for the treatment of anxiety, insomnia, and depression. About the size of a smart phone, the Alpha-Stim AID emits a mild electrical current via ear clip electrodes. The technical specifications for the Alpha-Stim® AID are shown on pages, 15-16. One-half of the devices will be active CES devices (0.5 Hz,  $100~\mu$ A (subsensory level), 50% duty cycle, biphasic asymmetrical rectangular waves) using ear clip electrodes. The other one-half of the devices (sham CES) will be identical to the active CES device except the ear clip electrodes will not emit electricity. The FDA has approved the device to be down classified from Class III to Class II (Federal Register, 2014). Subjects will complete a daily one hour CES treatment using ear clip electrodes (Figure 2.) with current set at fixed level of  $100~\mu$ A (subsensory level) for active CES treatment group for 6 weeks. The procedure will be the same for the sham group, but the Alpha-Stim® AID ear clips will not emit electricity.

Findings to date indicate that the Alpha-Stim® AID is an effective treatment with broad applications for a variety of syndromes for the management of anxiety, depression, and insomnia, or for the short-term relief of the symptoms of anxiety, depression and/or insomnia. In many cases it is the sole therapeutic method required.

#### Treatment Regimen:

The treatment regimen is one daily 60 minutes Alpha-Stim® CES treatment using ear clip electrodes for 6 weeks at 0.5 Hz. 50% duty cycle with a fixed current of  $100 \mu A$  (subsensory level). The sham CES unit is identical except the sham ear clip electrodes do not emit electricity.

Method for Assigning Subjects to Treatment Groups:

The blocked randomization method will be used to assign participants to active and sham groups (Efird, 2011). Participants will be assigned to CES treatment or sham CES using a 1:1 ratio. Electromedical Products International, Inc. (EPI) will randomize the assignment of appropriate devices to active or sham groups by using a random list of computer generated numbers (1 for active and 2 for sham) in randomly selected block sizes. An EPI device log will be developed as follows: The appropriate device, either active or sham will be assigned to a subject's number in the study (1 - 10, etc.), starting with number 1, in sequential order and the device's serial number will be listed on the EPI device log in the far-right column, Device Serial Number. The EPI log will remain in the EPI office. EPI will enter all device serial numbers on the Investigator device log in the order they are listed on the EPI device log. Study personnel will assign a device to a participant by using the next available device serial number in the order it is listed on the investigator device log. If a participant drops out of the study, that subject's device will be used for the replacement subject. If for some reason, the participant does not return the device, EPI will be notified and they will send the appropriate device, either active or sham, for the replacement subject. The device box will contain an equal number of active and sham CES device kits. The devices will be packed by EPI in the device box in the order of the device serial numbers on the device log. Only EPI has a list of numbers of the devices assigned to the active and sham groups. The PI, RA and participants are blinded to which participants have Alpha-Stim® CES active or sham devices until data analysis is complete. After the last participant completes the study and all data are entered, an individual completely independent of the study and data analysis, for example a database manager, will assign de-identified participants to unidentified groups using the serial numbers provided by EPI. After the completion of data analysis, blinding will be broken.

**D. Data Storage.** Describe how the data collected will be stored, location(s), how the confidentiality of individually identifiable information will be maintained (if applicable), and who will have access. (For audio and video recordings, include transcripts).

Privacy and confidentiality will be maintained for the participants during all study processes by keeping participant's materials in a sealed envelope prior to screening, assigning their names as numbers during questionnaire administration and to the treatment log. Initial screening and data collection will take place in a private clinic area designated by staff to maintain participant privacy and confidentiality. During recruitment potential participant's completed materials in a sealed envelope and place in a locked file cabinet in an inner-clinic office within the clinic to be picked by the PI or RA weekly. Hard copies of data will be stored in a locked file cabinet within an inner clinic office and then transported by the PI or RA to the PI's university office and locked in a file cabinet. For subsequent data collection, participants may also choose to complete study visits 1-3 during their current visit or at another designated location with the PI or RA. Numbers will be used in all written and digital records. No electronic data will be collected.

| <b>E. Records Retention.</b> For data collected, describe how records will be maintained, duration (minimum of three years), and responsible party. (For audio and video recordings, indicate time of destruction). |
|---|
| Only the PI and RA will have access to the actual names, addresses, and phone numbers of the participants. Contact information will be kept separate from participant data. This information will be secured in a locked cabinet in the PI's university office for a period of five years after data analysis at which time data will be destroyed. Paper data will be shredded |
| Risk to Participants; Mechanism of Protection; Outside Assistance |

A. Risk to Participants. Indicate the level of risk to participants.

| No risk | Y | | N | $\boxtimes$ |
|---|---|---|---|---|
| Minimal risk Definition: the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests. | Y | $\boxtimes$ | N | |
| Greater than minimal risk | Y | | N | $\boxtimes$ |

**B. Mechanism of Protection.** Describe **every potential risk** to human subjects that may result from participation in the research ("Risk"), and indicate the method or procedure to be used to mitigate the potential risk ("Protection Mechanism"). Consider physical, psychological, social, legal, and economic risks (e.g., breach of confidentiality, injury, psychological distress, pressure to conform, pressure to participate, etc).

| | Risk | Protection Mechanism |
|---|---|---|
| 1. | Breach of confidentiality | Confidentiality will be maintained for the participants by assigning their names as numbers during questionnaire administration and by assigning numbers to the treatment log. |
| 2. | Severe levels of anxiety or depression are identified | The PI or RA, who is an experienced clinicians, will make referrals to the appropriate resources and healthcare provider. |
| 3. | Side-effects: Side-effects seen in approximately 4,541 patients in controlled, open, uncontrolled conditions, and by physician survey and reasonably associated with the use of CES are dizziness (6 cases, 0.13%), skin irritation/electrode burns (5 cases, 0.11%), and headaches (9 cases, 0.20%). Prolonged CES treatment at higher than necessary currents may cause dizziness or nausea that can last from hours to days. | Side-effects are usually mild and self-limiting. Adverse effects are generally seen with treatment at higher than necessary currents. For this study, the active CES unit will be preset by the manufacturer and cannot be independently manipulated. Therefore, higher currents cannot occur. The sham CES unit will be inactive and the ear clip electrodes will not emit electricity. If side effects occur during the use of CES participants will be referred back to their OB/GYN. |
| 4. | As with any therapeutic intervention, not all participants in the treatment group will respond to the Alpha-Stim® AID. Participants randomly assigned to the SHAM group will not receive treatment. | PI or RA will discuss this possibility with participants during informed consent process. |
| 5. | | |
| 6. | | |
| 7. | | |
| 8. | | |
| 9. | В | |
| 10. | | |

C. Outside Assistance. If applicable, describe any outside assistance available to participants to mitigate the Risks stated above and how this information will be provided (e.g., medical care, counseling, etc).

This study is not expected to involve psychological, social, physical, economic, academic, or legal risks of harm to participants or living children any greater than those ordinarily encountered in daily life. However, if a participant is identified to have severe levels of stress, anxiety, or depression the PI or RA, who is an experienced clinicians, will make referrals to the appropriate resources and health care provider. If side effects occur during the use of CES participants will be referred back to their OB/GYN.

## Benefits to Participants; Benefits to Society

A. Benefits to Participants. If applicable, describe the potential benefits to participants as a result of taking part in the research (exclude payments/incentives). If there are no benefits, then state so.

Participants may benefit from this study by becoming more aware of their current mental health status and realizing perceptions about their own health and relationship to maternal functioning.

B. Benefits to Society. Describe the potential benefits to society or contribution to generalizable knowledge as a result of the research.

The information derived from this study can provide important information about the efficacy and adverse effects of a clinical interventions by controlling the variables that could impact the results of the study. It may also provide important information about maternal psychological distress that could translate to health care costs and use.

# Waiver of Informed Consent; Informed Consent Process

| A(1). Is a <u>waiver</u> of <u>signed</u> informed consent requested? (See Criteria for Waiver of Signed Informed Consent at the end of the HSRP for guidance). If "no," go to B. | Y 🗆 | N 🗵 | A(2). If <u>"yes,"</u> select which criteria applies, then go to B. (See Criteria for Waiver of Signed Informed Consent at the end of the HSRP for guidance). | I |
|---|---|---|---|---|
|---|---|---|---|---|

B. Informed Consent Process. Describe step-by-step how informed consent will be obtained from participants (i.e., who, what, where, when, how).

Note:

- 1) Participants must be given time to review the informed consent and supporting documents and ask questions.
- 2) For minor participants, researchers must obtain both parental informed consent and a separate child assent written at an appropriate reading
- 3) For participants whose first language is not English, informed consent may be required in English and non-English. In addition, submission of a Translator Certification or Interpreter Certification form may be required.

The potential participant will be notified if she qualifies for the study or does not meet the criteria for the study. If a new mother qualifies for the study, the PI or RA will briefly describe the study and time commitment. If the new mother agrees to participate, an appointment will be scheduled at the participants' next scheduled clinic visit or at the current time and location with the PI or RA to complete Visit 1. Participants may also choose to complete study visits 1-3 during their current visit or at another designated location with the PI or RA. The PI or RA will explain the study's purpose and procedures and read the consent form to all potential participants. After the potential participant's questions are addressed and verbal consent to participate is obtained, the new mother will sign the informed consent form.

# **Researcher Qualifications**

A. Describe qualifications or attach CVs/resumes for all personnel listed on the HSRP.

| The second of the second of th |
|---|
| See attached abbreviated CV (abbreviated) |
| ISee attached appreviated GV (appreviated) |
| Dec attached to the control of the c |

## Researcher Signatures

By signing this HSRP, the Researcher(s) certifies that he/she has read and understood the requirements and responsibilities set forth in the section entitled "Instructions and Researcher Certifications" in relation to the research. In addition, the Researcher (s) certifies that he/she will abide by any and all applicable federal, state, and/or institutional regulations, including any requirements from the Institutional Review Board (IRB) and/or the Office of Research Compliance (ORC).

| | Name | Conflict of Interest<br>(select one) | Date |
|-----------|------------|-------------------------------------------|------|
| PI | R | No conflict of interest with this project | |
| | Signature: | | |
| Co-PI (1) | | | |
| | Signature: | | |
| Co-PI (2) | * | | |
| | Signature: | | |
| Co-PI (3) | | | |
| | Signature: | | |
| Co-PI (4) | | | |
| | Signature: | | |
| Co-PI (5) | | | |
| | Signature: | | |

### **Determination of Level of Review**

The following research activities generally **do not** qualify for exempt review and will be reviewed at the level of expedited or full board:

- 1) Studies involving sensitive subject matters (e.g., abortion, AIDS/HIV, alcohol, body composition, criminal activity, drugs, depression, financial matters, learning disability, psychological well-being, sexual activity, suicide, etc).
- 2) Studies involving audiotaping and/or videotaping.

### **Exempt Review**

- 1) Research conducted in established or commonly accepted educational settings, involving normal education practices, such as (i.) research on regular and special education instructional strategies, or (ii.) research on the effectiveness of or the comparison among instructional techniques, curricula, or classroom management methods.
- 2) Research involving the use of educational tests (cognitive, diagnostic, aptitude, achievement), survey procedures, interview procedures or observation of public behavior, unless (i.) information obtained is recorded in such a manner that human subjects can be identified, directly or through identifiers linked to the subjects; and (ii.) any disclosure of human subjects' responses

- outside the research could reasonably place the subjects at risk of criminal or civil liability or be damaging to the subjects' financial standing, employability, or reputation.
- 3) Research involving the use of educational tests (cognitive, diagnostic, aptitude, achievement), survey procedures, interview procedures, or observation of public behavior that is not exempt under the previous paragraph, if (i.) the human subjects are elected or appointed public officials or candidates for public office; or (ii.) federal statute(s) require(s) without exception that the confidentiality of the personally identifiable information will be maintained throughout the research and thereafter.
- 4) Research involving the collection or study of existing data, documents, records, pathological specimens, or diagnostic specimens, if these sources are publicly available or if the information is recorded by the investigator in such a manner that subjects cannot be identified, directly or through identifiers linked to the subjects.
- 5) Research and demonstration projects that are conducted by or subject to the approval of federal department or agency heads, and that are designed to study, evaluate, or otherwise examine (i.) public benefit or service programs (ii.) procedures for obtaining benefits or services under these programs (iii.) possible changes in or alternatives to those programs or procedures; or (iv.) possible changes in methods or levels of payment for benefits or services under those programs
- 6) Taste and food quality evaluation and consumer acceptance studies (i.) if wholesome foods without additives are consumed or (ii.) if a food is consumed that contains a food ingredient at or below the level and for a use found to be safe, or agricultural chemical or environmental contaminant at or below the level found to be safe, by the Food and Drug Administration or approved by the Environmental Protection Agency or the Food Safety and Inspection Service of the U.S. Department of Agriculture

### **Expedited Review**

- (1) Clinical studies of drugs and medical devices only when condition (a) or (b) is met.
  - a. Research on drugs for which an investigational new drug application (21 CFR Part 312) is not required. (Note: Research on marketed drugs that significantly increases the risks or decreases the acceptability of the risks associated with the use of the product is not eligible for expedited review.)
  - b. Research on medical devices for which (i) an investigational device exemption application (21 CFR Part 812) is not required; or
     (ii) the medical device is cleared/approved for marketing and the medical device is being used in accordance with its cleared/approved labeling.
- (2) Collection of blood samples by finger stick, heel stick, ear stick, or venipuncture as follows:
  - a. from healthy, nonpregnant adults who weigh at least 110 pounds. For these subjects, the amounts drawn may not exceed 550 ml in an 8 week period and collection may not occur more frequently than 2 times per week; or
  - b. from other adults and children, considering the age, weight, and health of the subjects, the collection procedure, the amount of blood to be collected, and the frequency with which it will be collected. For these subjects, the amount drawn may not exceed the lesser of 50 ml or 3 ml per kg in an 8 week period and collection may not occur more frequently than 2 times per week.
- (3) Prospective collection of biological specimens for research purposes by noninvasive means.

  Examples: (a) hair and nail clippings in a nondisfiguring manner; (b) deciduous teeth at time of exfoliation or if routine patient care indicates a need for extraction; (c) permanent teeth if routine patient care indicates a need for extraction; (d) excreta and external secretions (including sweat); (e) uncannulated saliva collected either in an unstimulated fashion or stimulated by chewing gumbase or wax or by applying a dilute citric solution to the tongue; (f) placenta removed at delivery; (g) amniotic fluid obtained at the time of rupture of the membrane prior to or during labor; (h) supra- and subgingival dental plaque and calculus, provided the collection procedure is not more invasive than routine prophylactic scaling of the teeth and the process is accomplished in accordance with accepted prophylactic techniques; (i) mucosal and skin cells collected by buccal scraping or swab, skin swab, or mouth washings; (j) sputum collected after saline mist nebulization.
- (4) Collection of data through noninvasive procedures (not involving general anesthesia or sedation) routinely employed in clinical practice, excluding procedures involving x-rays or microwaves. Where medical devices are employed, they must be cleared/approved for marketing. (Studies intended to evaluate the safety and effectiveness of the medical device are not generally eligible for expedited review, including studies of cleared medical devices for new indications.)
  - Examples: (a) physical sensors that are applied either to the surface of the body or at a distance and do not involve input of significant amounts of energy into the subject or an invasion of the subject's privacy; (b) weighing or testing sensory acuity; (c) magnetic resonance imaging; (d) electrocardiography, electroencephalography, thermography, detection of naturally occurring radioactivity, electroretinography, ultrasound, diagnostic infrared imaging, doppler blood flow, and echocardiography; (e) moderate exercise, muscular strength testing, body composition assessment, and flexibility testing where appropriate given the

age, weight, and health of the individual.

- (5) Research involving materials (data, documents, records, or specimens) that have been collected, or will be collected solely for nonresearch purposes (such as medical treatment or diagnosis). (NOTE: Some research in this category may be exempt from the HHS regulations for the protection of human subjects. 45 CFR 46.101(b)(4). This listing refers only to research that is not exempt.)
- (6) Collection of data from voice, video, digital, or image recordings made for research purposes.
- (7) Research on individual or group characteristics or behavior (including, but not limited to, research on perception, cognition, motivation, identity, language, communication, cultural beliefs or practices, and social behavior) or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies. (NOTE: Some research in this category may be exempt from the HHS regulations for the protection of human subjects. 45 CFR 46.101(b) (2) and (b)(3). This listing refers only to research that is not exempt.)
- (8) Continuing review of research previously approved by the convened IRB as follows:
  - a. where (i) the research is permanently closed to the enrollment of new subjects; (ii) all subjects have completed all research related interventions; and (iii) the research remains active only for long-term follow-up of subjects; or
  - b. where no subjects have been enrolled and no additional risks have been identified; or
  - c. where the remaining research activities are limited to data analysis.
- (9) Continuing review of research, not conducted under an investigational new drug application or investigational device exemption where categories two (2) through eight (8) do not apply but the IRB has determined and documented at a convened meeting that the research involves no greater than minimal risk and no additional risks have been identified.

## **Criteria for Waiver of Signed Informed Consent**

- **(c)** An IRB may approve a consent procedure which does not include, or which alters, some or all of the elements of informed consent set forth above, or waive the requirement to obtain informed consent provided the IRB finds and documents that:
  - (1) The research or demonstration project is to be conducted by or subject to the approval of state or local government officials and is designed to study, evaluate, or otherwise examine: (i) public benefit or service programs; (ii) procedures for obtaining benefits or services under those programs; (iii) possible changes in or alternatives to those programs or procedures; or (iv) possible changes in methods or levels of payment for benefits or services under those programs; and
  - (2) The research could not practicably be carried out without the waiver or alteration.
- (d) An IRB may approve a consent procedure which does not include, or which alters, some or all of the elements of informed consent set forth in this section, or waive the requirements to obtain informed consent provided the IRB finds and documents that:
  - (1) The research involves no more than minimal risk to the subjects;
  - (2) The waiver or alteration will not adversely affect the rights and welfare of the subjects;
  - (3) The research could not practicably be carried out without the waiver or alteration; and
  - (4) Whenever appropriate, the subjects will be provided with additional pertinent information after participation.